CLINICAL TRIAL: NCT04316585
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of GSK2982772 in Participants With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Evaluate the Benefit and Safety of GSK2982772 in Moderate to Severe Psoriasis Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 208022
Record Dates: First submitted 2020-03-17; First posted 2020-03-20 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-08

CONDITIONS: Psoriasis
Keywords: Plaque Psoriasis; Modified Release; GSK2982772; Skin Biopsy
MeSH Terms: conditions — Psoriasis | interventions — GSK2982772

STUDY DESIGN:
Intervention Model Description: Participants will randomized in ratio of 2:1 to receive either 960 mg GSK2982772 or placebo
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study where sponsor will be unblinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants receiving GSK2982772 960 mg (Experimental): Participants will receive GSK2982772 960 mg oral tablets once daily for 12 weeks.
  Interventions: Drug: GSK2982772
- Participants receiving placebo (Placebo Comparator): Participants will receive GSK2982772 matching placebo oral tablets once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2982772 — GSK2982772 will be available as MR tablet at a unit dose strength of 480 mg.
  Arms: Participants receiving GSK2982772 960 mg
Drug: Placebo — GSK2982772 matching placebo tablets will be administered via the oral route.
  Arms: Participants receiving placebo

SUMMARY:
Plaque psoriasis is a chronic relapsing inflammatory skin disease that is characterized by keratinocyte hyper-proliferation and epidermal hyperplasia. Standard treatment for psoriasis generally requires long-term use of topical therapies, psoralen and ultraviolet A (PUVA), ultraviolet B (UVB) and/or systemic immunosuppressant therapies to achieve and maintain adequate disease control. This is a multicenter, randomized, double-blind study conducted in participants with moderate to severe plaque psoriasis. The study will evaluate the efficacy, safety, pharmacokinetic and pharmacodynamics profile of 960 milligram (mg) GSK2982772 administered as a once daily modified release (MR) formulation. Participants will be randomized in a 2:1 ratio to receive either 960 mg GSK2982772 or placebo for 12 weeks. The duration of the study, including Screening and follow-up, will be approximately 21 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Participants between 18 and 75 years of age inclusive, at the time of signing the informed consent.
* Diagnosis of plaque psoriasis for at least 6 months before Screening visit.
* Evidence of moderate to severe psoriasis, at Screening and Baseline before the first dose of study treatment, with: PASI score >=12; Psoriasis plaques involving BSA >=10 percent and sIGA>=3.
* Candidate for systemic therapy or phototherapy (includes naïve or previously treated), in the opinion of the Investigator.
* Agrees to avoid any prolonged exposure to natural or artificial sources of ultraviolet (UV) radiation from 28 days before Day 1 until the follow-up visit, which may potentially impact the participant's psoriasis in the opinion of the Investigator.
* Body mass index (BMI) within the range of 18.5 to 40.0 kilogram (kg)/meter square (m^2).
* Preclinical data has not identified risk of clinically relevant genotoxicity, however there is demonstrated/suspected risk of teratogenicity/fetotoxicity. Accordingly, the following contraceptive advice must be adhered to for male and female participants.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Male participants are eligible to participate if they agree to the following during the intervention period and for at least 2 days (i.e. 5 terminal half-lives of GSK2982772) after the last dose of study intervention: Refrain from donating sperm plus either: Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR Must agree to use contraception/barrier as detailed: Agree to use a male condom and will also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: Is not a WOCBP OR Is a WOCBP and using a contraceptive method that is highly effective preferably with low user dependency, during the intervention period and for at least 28 days (i.e. until resolution of potential drug interaction with combined hormonal contraceptives) after the last dose of study intervention. The Investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention. A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 24 hours before the first dose of study intervention. If a urine test cannot be confirmed as negative (example an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
* The Investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and protocol.

Exclusion Criteria:

* Non-plaque forms of psoriasis (example erythrodermic, guttate, or pustular), in the opinion of the Investigator.
* Drug-induced psoriasis (example a new onset of psoriasis or an exacerbation from beta blockers, calcium channel blockers, lithium or anti-Tumor-Necrosis Factor [TNF] therapies).
* Diagnosis of psoriatic arthritis, uveitis, inflammatory bowel disease, or other immune-mediated conditions that are commonly associated with psoriasis for which a participant requires current systemic (oral, subcutaneous [SC], or intravenous [IV]) (including corticosteroids and biologics) immunosuppressant medical treatment.
* Current Suicidal Ideation Behavior (SIB) as measured using the Columbia Suicide Severity Rating Scale (C-SSRS) or a history of attempted suicide at Screening and before first dose of study treatment.
* Active infection, or a history of infections as follows: Hospitalization for treatment of infection within 60 days before Day 1; Current use of any suppressive therapy for a chronic infection (such as pneumocystis jirovecii, cytomegalovirus, herpes simplex virus, herpes zoster virus and atypical mycobacteria); Use of parenteral (IV or intramuscular) antibiotics (anti-bacterials, antivirals, antifungals, or anti-parasitic agents) within 60 days before Day 1; History of opportunistic infections within 1 year of Screening (example pneumocystis jirovecii, Cytomegalovirus [CMV] pneumonitis, aspergillosis). This does not include infections that may occur in immunocompetent individuals, such as fungal nail infections or vaginal candidiasis, unless it is of an unusual severity or recurrent nature; History of recurrent, chronic or other active infection that in the opinion of the Investigator may put the participant at unacceptable risk or interfere/confound the integrity of study data; Positive test for Severe Acute Respiratory Syndrome-Related Coronavirus 2 (SARS-CoV-2) at screening or interaction with known Coronovirus Disease 2019 (COVID19) positive contacts within 14 days prior to Day 1; History of latent or active Tuberculosis (TB), irrespective of treatment status; A positive diagnostic TB test at Screening defined as a positive QuantiFERON-TB Gold plus test.
* Current or history of liver disease, known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Current or history of renal disease.
* Significant unstable or uncontrolled cardiovascular disease including uncontrolled hypertension.
* Hereditary or acquired immunodeficiency disorder, including immunoglobulin deficiency.
* History of major organ transplant (example heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant.
* Planned surgical procedure that makes the participant unsuitable for the study, in the opinion of the Investigator.
* History of malignant neoplasm within the last 5 years, except for adequately treated cancers of the skin (basal or squamous cell carcinoma) or carcinoma in situ of the uterine cervix that has been fully treated and shows no evidence of recurrence after at least 12 months following treatment.
* History of significant progressive neurologic disorders including, but not limited to, progressive Multiple Sclerosis (MS), Amyotrophic Lateral Sclerosis (ALS), Alzheimer's and dementia.
* History of a medical condition other than plaque psoriasis, or other considerations, which may confound interpretation of efficacy or safety study data, or put the participant at unacceptable risk, in the opinion of the Investigator.
* History of lack of primary response to anti-TNF biologic therapies (either approved or experimental) at approved doses (or at the doses received if experimental therapies) after at least 3 months of therapy.
* Participant has previous exposure to 3 or more biologic therapies of any mechanism of action.
* Treatment with the prohibited therapies or changes to those treatments, within the specified timeframe. Other medications (including vitamins, herbal and dietary supplements) will be considered on a case-by-case basis and will be allowed if the medication will not interfere with the study procedures or compromise participant safety, in the opinion of the Investigator.
* Participation in a clinical trial and has received an investigational product within 30 days or 5 half-lives whichever is longer (or 12 weeks for biologic therapies), before the first dose of study medication, or plans to take part in another clinical trial at the same time as participating in this clinical trial.
* Exposure to more than four investigational products within 12 months prior to the first dosing day.
* Average QT Duration Corrected for Heart Rate (QTc) >450 milliseconds (msec) or QTc>480 msec in participants with bundle branch block at Screening and before first dose of study treatment. The QTc is the QT interval corrected for heart rate according to Fridericia's formula (QTcF). It is either machine-read or manually over-read.
* Alanine transferase (ALT) >2 × upper limit of normal (ULN)
* Bilirubin >1.5 × ULN at Screening (isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Estimated glomerular filtration rate (GFR) by Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI) <60 milliliter (mL)/minute (min)/1.73 m^2.
* Hemoglobin < 10 gram per deciliter (g/dL); hematocrit < 30 percent, white blood cell count <= 3000 /cubic millimeter (mm^3) (<= 3.0 x 10^9/Liter); platelet count <= 100,000 /microliter (μL) (<= 100 x 10^9/Liter); absolute neutrophil count (<= 1.5 x 10^9/Liter).
* Presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb).
* Presence of hepatitis C antibody at Screening. Participants with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative hepatitis C Ribonucleic acid (RNA) test is obtained.
* Positive serology for Human Immunodeficiency Virus (HIV) 1 or 2.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 3 months.
* History of alcohol or drug abuse, that would interfere with the ability to comply with the study or interfere with interpretation of the study, in the opinion of the Investigator.
* History of sensitivity to any of the study treatments, or components thereof, or a history of drug or other allergy that contraindicates their participation (including lidocaine or other local anesthetic), in the opinion of the Investigator or Medical Monitor.
* History of receiving a live or attenuated vaccine within 30 days of randomization OR plan to receive a live or attenuated vaccination during the study until completion of the follow-up visit.
* History of hypertrophic or keloid scarring.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Canada (7):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Oakville, Ontario
  - GSK Investigational Site, Peterborough, Ontario
  - GSK Investigational Site, Québec, Quebec
- GSK Investigational Site, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 39 participants were screened, of which 29 participants were enrolled in the study.
Groups:
- GSK2982772 960 mg: Participants received GSK2982772 960 mg oral tablets once daily for 12 weeks.
- Placebo: Participants received GSK2982772 matching placebo oral tablets once daily for 12 weeks.
Period: Overall Study
Arm/Group | GSK2982772 960 mg | Placebo
Started | 19 | 10
Completed | 13 | 5
Not Completed | 6 | 5
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3
Not completed — SUBJECT REACHED PROTOCOL-DEFINED STOPPING CRITERIA | 0 | 1
Not completed — INVESTIGATOR DISCRETION | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2982772 960 mg | Placebo | Total
Number analyzed (Participants) | 19 | 10 | 29
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 50.1 (15.97) | 46.5 (12.52) | 48.8 (14.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 16 | 5 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - South East Asian Heritage | 1 | 0 | 1
  Mixed White race | 0 | 1 | 1
  Mixed race | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 17 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage (%) of Participants Who Achieved Greater Than or Equal (>=) to 75% Improvement From Baseline in Psoriasis Area Severity Index (PASI) Score at Week 12
Description: The Psoriasis area severity index (PASI) is a standard tool for assessing the severity of psoriasis that considers the overall severity of erythema, induration, and scaling (each scored separately), and the extent of body surface area (BSA) affected with psoriasis. The 3 clinical signs are each graded on a 5-point scale (0=none to 4=severe) and the percent BSA affected is scored on a 7-point scale (0= 0% skin with psoriasis to 6= ≥ 90% skin with psoriasis). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. The PASI is a composite scoring assessed by the investigator for the severity of lesions and the area affected into a single score with a range of 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Note: The 95% credible interval (CrI) was reported as a method of dispersion.
Time Frame: Baseline and Week 12
Population: The analysis was performed on the Intent to Treat Set that includes all participants who were randomized to study intervention in the study and who received at least one dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | GSK2982772 960 mg | Placebo
Number analyzed (Participants) | 19 | 10
Percentage of Participants | 5 [0.4 to 21] | 0 [0 to 18.2]
Statistical Analysis 1: Comparison: GSK2982772 960 mg vs Placebo; Bayesian logistic regression. An informative prior was used for the placebo response in this statistical analysis, the prior for placebo response rate was of the form: 90% weight on Be (5.39, 69) and 10% on Be (1/3,1/3). The prior was derived from historical data from similar clinical trials using meta-analytic predictive prior (MAP) approach. All other parameters took vague priors; Test type: Superiority; Bayesian Logistic Regression Model; The model was adjusted for treatment (GSK2982772 vs placebo), baseline PASI score and prior biologic use (yes/no); Mean Difference (Final Values) = -2.28, 95% CI 2-sided [-9.19 to 8.28] — Posterior median and 95% CrI for the true difference in proportion of responders (GSK2982772 - placebo)
Statistical Analysis 2: Comparison: GSK2982772 960 mg vs Placebo; Test type: Superiority; Bayesian Logistic Regression Model; The model was adjusted for treatment (GSK2982772 vs placebo), baseline PASI score and prior biologic use (yes/no); Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-4.81 to 8.07] — Posterior median and 95% CrI for the true difference in proportion of responders (GSK2982772 - placebo)

2. Secondary Outcome: Percentage of Participants Who Achieved >=50% Improvement From Baseline in Psoriasis Area Severity Index (PASI) Score at Week 12
Description: The PASI is a standard tool for assessing the severity of psoriasis that considers the overall severity of erythema, induration, and scaling (each scored separately), and the extent of body surface area (BSA) affected with psoriasis. The 3 clinical signs are each graded on a 5-point scale (0=none to 4=severe) and the percent BSA affected is scored on a 7-point scale (0= 0% skin with psoriasis to 6= ≥ 90% skin with psoriasis). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. The PASI is a composite scoring assessed by the investigator for the severity of lesions and the area affected into a single score with a range of 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Note: The 95% CrI was reported as a method of dispersion.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | GSK2982772 960 mg | Placebo
Number analyzed (Participants) | 19 | 10
Percentage of Participants | 42 [22.1 to 64.2] | 20 [3.9 to 49.7]

3. Secondary Outcome: Percentage of Participants Who Achieved >=90% Improvement From Baseline in Psoriasis Area Severity Index (PASI) Score at Week 12
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | GSK2982772 960 mg | Placebo
Number analyzed (Participants) | 19 | 10
Percentage of Participants | 0 [0 to 10.1] | 0 [0 to 18.2]

4. Secondary Outcome: Percentage of Participants Who Achieved >=100% Improvement From Baseline in Psoriasis Area Severity Index (PASI) Score at Week 12
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | GSK2982772 960 mg | Placebo
Number analyzed (Participants) | 19 | 10
Percentage of Participants | 0 [0 to 10.1] | 0 [0 to 18.2]

5. Secondary Outcome: Change From Baseline in Psoriasis Area Severity Index (PASI) Scores at Week 12
Description: The PASI is a standard tool for assessing the severity of psoriasis that considers the overall severity of erythema, induration, and scaling (each scored separately), and the extent of body surface area (BSA) affected with psoriasis. The 3 clinical signs are each graded on a 5-point scale (0=none to 4=severe) and the percent BSA affected is scored on a 7-point scale (0= 0% skin with psoriasis to 6= ≥ 90% skin with psoriasis). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. The PASI is a composite scoring assessed by the investigator for the severity of lesions and the area affected into a single score with a range of 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | GSK2982772 960 mg | Placebo
Number analyzed (Participants) | 19 | 10
Scores on a Scale | -8.82 (4.501) | -6.98 (5.228)

6. Secondary Outcome: Percentage of Participants Who Have a Static Investigator's Global Assessment (sIGA) Score of 0 or 1 at Week 12
Description: Either investigator or his designee completed a global assessment of disease activity using the physician global assessment item. A 5-point scoring system was used to measure the severity of psoriatic lesions over the entire body at the time of evaluation. The 5-point scoring system ranging from 0 to 4 where 0 = Clear, 1 = Almost Clear, 2 = Mild, 3 = Moderate and 4=Severe. Percentage of participants who have a sIGA score of 0=clear or 1=almost clear at Week 12 was summarized. Note: The 95% CrI was reported as a method of dispersion.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | GSK2982772 960 mg | Placebo
Number analyzed (Participants) | 19 | 10
Percentage of Participants | 11 [1.9 to 28.9] | 0 [0 to 18.2]

7. Secondary Outcome: Change From Baseline in Psoriatic Body Surface Area (BSA) at Week 12
Description: The BSA affected with psoriasis was evaluated at all study visits by the Investigator or suitably trained delegate. As a reference, the area of the whole palm was counted as 1% BSA. Change from Baseline was calculated as Post-Baseline visit values minus Baseline value.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Body Surface Area
Arm/Group | GSK2982772 960 mg | Placebo
Number analyzed (Participants) | 19 | 10
Percentage of Body Surface Area | -5.2 (6.30) | -3.7 (4.41)

8. Secondary Outcome: Number of Participants With Any Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Time Frame: Up to Day 120
Population: The analysis was performed on the Safety Set that included all participants in the enrolled population who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2982772 960 mg | Placebo
Number analyzed (Participants) | 19 | 10
Participants | 12 | 6

9. Secondary Outcome: Number of Participants With Drug Related AEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. The investigator was obligated to assess the relationship between study intervention and each occurrence of each AE.
Time Frame: Up to Day 120
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2982772 960 mg | Placebo
Number analyzed (Participants) | 19 | 10
Participants | 5 | 4

10. Secondary Outcome: Number of Participants With Common (Occurring at Least 5%) Non Serious AEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Non serious AEs are AEs that are not Serious Adverse Events (SAEs). All AEs occurring at least 5% in either arm were reported. Note: As both arms had small sample sizes, single occurrences of an AE met the 5% threshold for reporting.
Time Frame: Up to Day 120
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2982772 960 mg | Placebo
Number analyzed (Participants) | 19 | 10
Participants
  Neutropenia | 1 | 0
  Tinnitus | 1 | 0
  Dry eye | 1 | 0
  Diarrhea | 1 | 1
  Allergy to arthropod sting | 1 | 0
  Herpes zoster | 1 | 0
  Alanine aminotransferase increased | 0 | 1
  Aspartate aminotransferase increased | 0 | 1
  Blood creatinine abnormal | 1 | 0
  Creatinine renal clearance abnormal | 2 | 0
  Hepatitis E antibody positive | 0 | 1
  Neutrophil count decreased | 1 | 0
  White blood cell count decreased | 1 | 0
  Back pain | 2 | 1
  Headache | 3 | 3
  Suicidal ideation | 0 | 1
  Nasal congestion | 0 | 1
  Intertrigo | 0 | 1
  Pruritus | 0 | 1
  Psoriasis | 1 | 0
  Rash | 0 | 1
  Hypertension | 0 | 1

11. Secondary Outcome: Number of Participants With AEs Leading to Permanent Discontinuation of Study Intervention
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. All AEs which led to discontinuation of the study drug were reported.
Time Frame: Up to Day 120
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2982772 960 mg | Placebo
Number analyzed (Participants) | 19 | 10
Participants | 2 | 2

12. Secondary Outcome: Number of Participants With SAEs Including Any SAEs, SAEs Related to Study Intervention, and Fatal SAEs
Description: An SAE is defined as any untoward medical occurrence that, at any dose, results in death, was life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect and other situations according to medical or scientific judgement. All SAEs, SAEs related to the study drug, and fatal SAEs were reported.
Time Frame: Up to Day 120
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2982772 960 mg | Placebo
Number analyzed (Participants) | 19 | 10
Participants
  All SAEs | 1 | 0
  Study drug related SAE | 1 | 0
  Fatal SAE | 0 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, SAEs and non-serious AEs were collected from the start of study treatment including the Follow-up visit up to Day 120.
Description: All AEs and SAEs were reported for the Safety Population which comprised of all participants in the enrolled population who received at least one dose of study intervention.
Arm/Group | GSK2982772 960 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/10
Other Adverse Events (participants affected / at risk) | 11/19 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2982772 960 mg (N=19) | Placebo (N=10)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2982772 960 mg (N=19) | Placebo (N=10)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine abnormal (Investigations) | 1 (1) | 0 (0)
Creatinine renal clearance abnormal (Investigations) | 2 (2) | 0 (0)
Hepatitis E antibody positive (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 3 (6)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT04316585/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT04316585/SAP_001.pdf